CLINICAL TRIAL: NCT00869440
Title: A Phase IIa, Randomized, Controlled, Double-Blind, Dose-Finding Study Evaluating the Safety and Pharmacodynamics of CNS 7056 in Patients Undergoing Diagnostic Upper GI Endoscopy
Brief Title: Dose-Finding Safety Study Evaluating Remimazolam (CNS 7056) in Patients Undergoing Diagnostic Upper GI Endoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS 7056-003
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Procedural Sedation; Endoscopy
Keywords: CNS 7056; Procedural Sedation; Sedation; Endoscopy
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1: Remimazolam (CNS 7056) 0.10 mg/kg (Experimental): Remimazolam (CNS 7056) 0.10 mg/kg iv
  Interventions: Drug: CNS 7056
- 2: Remimazolam (CNS 7056) 0.15 mg/kg (Experimental): Remimazolam (CNS 7056) 0.15 mg/kg iv
  Interventions: Drug: CNS 7056
- 3: Remimazolam (CNS 7056) 0.20 mg/kg (Experimental): Remimazolam (CNS 7056) 0.20 mg/kg iv
  Interventions: Drug: CNS 7056
- 4: Midazolam 0.075 mg/kg (Experimental): Midazolam 0.075 mg/kg iv
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: CNS 7056 — Administered as a single intravenous injection by a syringe driver over 1 minute
  Other Names: remimazolam
  Arms: 1: Remimazolam (CNS 7056) 0.10 mg/kg; 2: Remimazolam (CNS 7056) 0.15 mg/kg; 3: Remimazolam (CNS 7056) 0.20 mg/kg
Drug: Midazolam — Administered as a single intravenous injection by a syringe driver over 1 minute
  Other Names: Versed
  Arms: 4: Midazolam 0.075 mg/kg

SUMMARY:
The purpose of this study was to assess the safety and efficacy of CNS 7056 as a procedural sedative at three dose levels compared to midazolam during a diagnostic upper GI endoscopy.

DETAILED DESCRIPTION:
This was a randomized, double-blind, parallel-group, dose-finding study assessing the safety and efficacy of three dose levels of CNS 7056 compared with midazolam in patients undergoing diagnostic upper GI endoscopy.

Patients who met all study entry criteria and completed screening procedures were randomly assigned to 1 of 4 treatment groups: CNS 7056 0.10 mg/kg,0.15 mg/kg, or 0.20 mg/kg; or midazolam 0.075 mg/kg. Patients received their assigned treatment administered as a single intravenous injection by a syringe driver over 1 minute. The endoscopy started when a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score of ≤3 has been reached, but no earlier than 90 seconds after Time 0 (the start of study drug injection). Rescue with sedative medication (midazolam 1-2 mg) was be permitted at the discretion of the administering physician.

Efficacy assessments consisted of the MOAA/S scores, Aldrete scores, and drowsiness measures using a Visual Analogue Scale (VAS). Cognitive function was assessed by the Hopkins Verbal Learning Test-Revised™ (HVLT-R™) and memory for the procedure by the Brice Questionnaire.

Safety assessments included adverse events, physical examinations, vital signs, ECGs, pulse oximetry measurements, clinical laboratory tests, and pain on injection using a VAS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18 to 65 years inclusive, scheduled to undergo diagnostic upper GI endoscopy.
* American Society of Anesthesiologists Physical Status (ASA PS) Score I or II.
* Weight range 60 to 120 kg inclusive.
* Body mass index (BMI) 18 to < 30 kg/m2.
* Patients with no clinically significant abnormalities in 12 lead ECG recorded at Screening.
* Female with a negative serum human chorionic gonadotropin (hCG) pregnancy test result at Screening and negative urine hCG pregnancy test result on Day 1 before the endoscopy procedure.
* Patients with negative drugs of abuse serum result at Screening and negative drugs of abuse urine result on Day 1 before the endoscopy procedure.
* Patient has a negative serum ethanol test result at Screening and a negative ethanol saliva test result on Day 1 before the endoscopy procedure.
* Patient voluntarily signs and dates an informed consent form (ICF) that is approved by an investigational review board (IRB) prior to the conduct of any study procedure.
* Patient is willing and able to comply with study requirements and return for a Follow up Visit (Visit 3 ± 1 day) after the endoscopy procedure.

Exclusion Criteria:

* Patients with a suspected upper GI bleed an conditions predisposing to hemorrhage at the discretion of the investigator.
* Has a known sensitivity to benzodiazepines, flumazenil, or anesthetic agents, or a medical condition such that these agents are contraindicated.
* Patients with evidence of uncontrolled renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction, in the opinion of the investigator or medical monitor.
* Patients taking an agent that inhibits cytochrome P450 subtype 3A4 (CYP3A4) or patients who have taken such an agent within 14 days prior to study start or within the duration of 7 half lives of the drug, whichever is longer.
* Patients in receipt of any investigational drug within 30 days or less than 7 half lives (whichever is longer) before the start of the study, or scheduled to receive one during the study period.
* Chronic use of benzodiazepines for any indication (eg, insomnia, anxiety, spasticity).
* Has known or suspected history of alcoholism or drug abuse or misuse within 2 years of Screening or evidence of tolerance or physical dependence before dosing with study drug.
* Patients with clinically significant findings at Screening that, in the investigator's opinion, should exclude them from the study.
* Patients with a history of laboratory results that show the presence of hepatitis B surface antigen (HBs Ag), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV).
* Patients with an inability to communicate well in English with the investigator.
* Lactating female patients.
* Patients in whom management of airway is judged to be difficult due to:

  * obesity (weight > 120 kg, or BMI ≥ 30 kg/m2),
  * thyro mental distance ≤ 4 cm ("short neck"), or
  * Mallampati score of 4 (Appendix IV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Helen Keller Hospital, Sheffield, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Miami Research Associates, South Miami, Florida
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Charlottesville Medical Research, Charlottesville, Virginia

REFERENCES:
- [Result] Borkett KM, Riff DS, Schwartz HI, Winkle PJ, Pambianco DJ, Lees JP, Wilhelm-Ogunbiyi K. A Phase IIa, randomized, double-blind study of remimazolam (CNS 7056) versus midazolam for sedation in upper gastrointestinal endoscopy. Anesth Analg. 2015 Apr;120(4):771-80. doi: 10.1213/ANE.0000000000000548. PMID 25502841

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: CNS 7056 0.10 mg/kg; 2: CNS 7056 0.15 mg/kg; 3: CNS 7056 0.20 mg/kg: CNS 7056: Administered as a single intravenous injection by a syringe driver over 1 minute
Period: Overall Study
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg
Started | 25 | 25 | 25 | 25
Completed | 23 | 24 | 25 | 25
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (13.33) | 38.8 (14.08) | 43.2 (13.95) | 44.6 (13.64) | 41.1 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 16 | 12 | 54
  Male | 12 | 12 | 9 | 13 | 46
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 100
Height [Mean (Standard Deviation); unit: cm] | 169.33 (9.603) | 168.42 (10.283) | 168.97 (7.432) | 171.55 (9.650) | 169.57 (9.241)
Weight [Mean (Standard Deviation); unit: kg] | 73.22 (10.583) | 75.17 (10.869) | 75.13 (11.027) | 75.45 (10.099) | 74.74 (10.526)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 25.47 (2.091) | 26.43 (2.158) | 26.24 (2.725) | 25.59 (2.262) | 25.93 (2.324)

OUTCOME MEASURES:

1. Primary Outcome: Success Rates of the Procedure
Description: Success of the procedure is a composite endpoint consisting of: MOAA/S scores ≤4 on three consecutive measurements after administration of study drug AND completion of the endoscopy procedure AND no requirement for rescue sedative medication AND no requirement for manual or mechanical ventilation
Time Frame: From start of study drug injection to patient discharge
Population: All randomized patients who received a dose of study drug, underwent the endoscopy procedure, and had at least 1 efficacy assessment (Intent-to-treat population)
Measure: Count of Participants; unit: Participants
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg
Number analyzed (Participants) | 25 | 25 | 25 | 25
Participants | 8 | 14 | 16 | 11

2. Secondary Outcome: Time to Fully Alert
Description: Time to first of 3 consecutive Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores of 5 following study drug administration in patients who underwent the endoscopy procedure
Time Frame: From study drug administration until fully alert criteria are reached
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg
Number analyzed (Participants) | 25 | 25 | 25 | 25
minutes | 11 (10.04) | 13.4 (6.51) | 12.1 (5.26) | 17.2 (16.71)

3. Secondary Outcome: Time to Ready for Discharge
Description: Time to first of 3 consecutive Aldrete scores ≥9 after the end endoscopy procedure
Time Frame: From the end of the endoscopy procedure up to 120 minutes or until 3 consecutive Aldrete scores of ≥9 are reached, whichever occurs first
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg
Number analyzed (Participants) | 25 | 25 | 25 | 25
minutes | 14 (9.96) | 12.8 (5.96) | 11.8 (4.96) | 17.2 (12.81)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Time 0 on Day 1 to the Follow-up Visit on Day 4, and were followed until resolution (with or without sequelae) up to a maximum of 30 days after Time 0.
Description: Total number of participants affected with Other (Not Including Serious) Adverse Events represents overall number of participants with non-serious TEAEs reported with a threshold of 5% in any of the arms
Arm/Group | 1: CNS 7056 0.10 mg/kg | 2: CNS 7056 0.15 mg/kg | 3: CNS 7056 0.20 mg/kg | 4: Midazolam 0.075 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 8/25 | 9/25 | 10/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1: CNS 7056 0.10 mg/kg (N=25) | 2: CNS 7056 0.15 mg/kg (N=25) | 3: CNS 7056 0.20 mg/kg (N=25) | 4: Midazolam 0.075 mg/kg (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 4 | 5 | 6 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 2 | 2
Pharyngeolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submission for publication, presentation or use, sponsor shall review and comment any proposed oral or written publication, which period may be extended for an additional 30 days. To seek patent protection, sponsor shall have the right to delay the proposed publication for an additional 60 days.